CLINICAL TRIAL: NCT04271111
Title: Computerized Intervention for Interpersonal Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Brittany Mathes, Graduate Student, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.26213
Record Dates: First submitted 2019-03-25; First posted 2020-02-17 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Hostility

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into active treatment or control condition.
Who Masked: Participant
Masking Description: Participants will not know what condition they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Computerized intervention aimed at reducing perceived hostility.
  Interventions: Behavioral: Online Treatment for Interpersonal Stress
- Control condition (Active Comparator): Computerized intervention aimed at increasing overall physical health.
  Interventions: Behavioral: Physical Health Education Tool

INTERVENTIONS:
Behavioral: Online Treatment for Interpersonal Stress — Intervention designed to build social support and reduce loneliness by giving participants skills to strengthen their relationships
  Arms: Active treatment
Behavioral: Physical Health Education Tool — Intervention designed to improve physical health through exercise, eating habits, and sleep
  Arms: Control condition

SUMMARY:
This study assesses whether a computerized intervention can be used to decrease perceived hostility in hostile individuals.

DETAILED DESCRIPTION:
This study will investigate whether a brief computerized intervention can decrease perceived hostility of interpersonal situations. Participants will be randomized into an active treatment or control condition. We hypothesize that participants in the treatment condition will have lower perceived hostility at post treatment than those in the waitlist condition.

ELIGIBILITY:
Inclusion Criteria:

* Increased hostility based on the Buss Perry Aggression Questionnaire

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in Cook Medley Hostility Inventory | Baseline, one hour, one week, one month
  Self-report measure assessing hostility using a true/false scale with higher scores indicating higher levels of hostility.
Changes in Word Sentence Association Paradigm-Hostility | Baseline, one hour, one week, one month
  Self-report measure assessing hostility using a 6-point scale with higher scores indicating higher levels of hostile interpretation bias.
Changes in Alcohol Use Disorders Identification Test | Baseline, one hour, one week, one month
  Self-report measure assessing symptoms of alcohol use disorder with higher scores indicating more severe symptoms.
Changes in Drinking Motives Questionnaires | Baseline, one hour, one week, one month
  Self-report measure assessing motives for drinking, including social, recreational, and coping. Higher scores indicate greater likelihood of drinking for each motive.
Changes in alcohol use | Baseline, one hour, one week, one month
  Participants will provide the number of standard drinks of alcohol they drank each day in the past month.

SECONDARY OUTCOMES:
Changes in Self Stigma of Seeking Help | Baseline, one hour, one week, one month
  Self-report measure assessing stigma associated with seeking help for psychological problems. Higher scores indicate greater negative attitudes toward psychosocial treatment.
Changes in Perceived Stigma and Barriers to Care for Psychological Treatment | Baseline, one hour, one week, one month
  Self-report measure assessing stigma associated with seeking help for psychological problems. Higher scores indicate greater negative attitudes toward psychosocial treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No